CLINICAL TRIAL: NCT01711827
Title: A Phase 1, Open-label, Sequential Study of the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Prednisone in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Prednisone in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0024
Record Dates: First submitted 2012-10-19; First posted 2012-10-22 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Subjects; Pharmacokinetics of Isavuconazole; Pharmacokinetics of Prednisolone
Keywords: isavuconazole; prednisone; prednisolone; BAL8557; healthy volunteers
MeSH Terms: interventions — isavuconazole; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and Prednisone (Experimental): Single dose of prednisone on Days 1 and 9, isavuconazole 3 times a day (TID) on Days 5-6, isavuconazole once a day (QD) on Days 7-10
  Interventions: Drug: Isavuconazole; Drug: Prednisone

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL8557
Drug: Prednisone — oral

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of prednisolone after single dose administration of prednisone. This study will also assess the safety and tolerability of isavuconazole alone and in combination with prednisone.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* Results for aspartate aminotransferase (ALT) must be ≤ upper limit of normal and total bilirubin must be ≤ 1.5 mg/dL
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death or a close relative at a young age due to possible or probably cardiac causes
* The subject has a history of tuberculosis or exposure to anyone known or suspected to have tuberculosis or any illness that might confound the results of the study or pose additional risk in administering study drug to the subject
* The subject has a positive result for hepatitis C antibodies, hepatitis B surface antigen, or QuantiFERON®-TB Gold test at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products including prednisone or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse or a positive drug and/or alcohol screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of plasma prednisolone: AUClast, | Predose on Days 1 and 9 and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (Days 2 and 10), and 48 (Days 3 and 11) hours postdose
  Area under the concentration-time curve (AUC) from the time of dosing to the last quantifiable concentration (AUC last)
Pharmacokinetics of plasma prednisolone: AUCinf | Predose on Days 1 and 9 and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (Days 2 and 10), and 48 (Days 3 and 11) hours postdose
  AUC from the time of dosing to infinity (AUCinf),
Pharmacokinetics of plasma prednisolone: Cmax | Predose on Days 1 and 9 and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (Days 2 and 10), and 48 (Days 3 and 11) hours postdose
  Maximum concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics of plasma isavuconazole concentration: Trough concentration (Ctrough) | Day 7 predose; Day10 predose and Day 11 postdose
Composite of pharmacokinetics of plasma isavuconazole concentration: AUCtau, Cmax, and tmax | Day 8 predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 16 hours postdose; Day 9 predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 hours postdose
  AUC during the time interval between consecutive dosing (AUCtau), Cmax, and time to attain Cmax (tmax)
Composite of pharmacokinetics of plasma prednisone: AUClast, AUCinf, Cmax, tmax, t1/2, Vz/F, and CL/F | Predose on Days 1 and 9 and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (Days 2 and 10), and 48 (Days 3 and 11) hours postdose
  Apparent terminal elimination half life ( t1/2), apparent volume of distribution (Vz/F), and apparent body clearance after oral dosing (CL/F)
Composite of pharmacokinetics of plasma prednisolone: t max and t1/2 | Predose on Days 1 and 9 and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (Days 2 and 10), and 48 (Days 3 and 11) hours postdose
Safety assessed by recording of adverse events, laboratory evaluations, electrocardiograms (ECGs) and vital signs | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel International, LLC, Glendale, California, United States